CLINICAL TRIAL: NCT07278700
Title: The Fever Clinic Acute Respiratory Cohort (FACTS): A Prospective Real-World Cohort Study of Patients Presenting to Fever Clinics: Clinical Features, Laboratory and Radiographic Findings, and Long-Term Outcomes of Acute Respiratory Infections
Brief Title: The Fever Clinic Acute Respiratory Cohort
Acronym: FACTS
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Huadong Hospital (Other)
Responsible Party: Principal Investigator, Zhijun Bao, President, Fudan University
Other Study IDs: FACTS
Record Dates: First submitted 2025-11-24; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Infections; Febrile Illnesses; Community-acquired Pneumonia; Viral Respiratory Tract Infections; Influenza-like Illness
Keywords: Respiratory Tract Infections; Fever; Community-Acquired Pneumonia; Anti-Bacterial Agents; Disease Progression
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Tract Infections; Fever; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pneumonia Cohort
  Interventions: Other: No intervention involved
- Non-Pneumonia Cohort
  Interventions: Other: No intervention involved

INTERVENTIONS:
Other: No intervention involved — This is a observational study so no intervention involved.

SUMMARY:
This prospective cohort study aims to characterize the natural progression and outcomes of acute respiratory infections among patients presenting to fever clinics. At enrollment, patients' clinical symptoms, laboratory findings, and chest imaging data will be collected. Longitudinal follow-up will be conducted to evaluate disease progression, complications, and long-term outcomes.

As an observational study, no interventions are involved; all patients receive routine clinical management as directed by their attending physicians. This real-world study design enables the assessment of the natural course of acute respiratory infections and the identification of factors associated with clinical outcomes.

DETAILED DESCRIPTION:
This prospective cohort study aims to characterize the natural history and outcomes of acute respiratory infection in patients presenting to fever clinics. Upon enrollment, patients' clinical symptoms, laboratory parameters, and chest imaging data will be collected. Subsequent longitudinal follow-up will be performed to assess disease progression, complications, and long-term outcomes.

As an observational study, no interventions are implemented; all patients receive standard-of-care management as determined by their attending physicians. This real-world study design allows for the evaluation of the natural progression of acute respiratory infections and the identification of factors associated with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (based on official identification document).
* Presence of fever at the time of visit or within 24 hours prior to the visit, defined as a documented temperature of ≥37.3°C axillary/tympanic, ≥37.8°C orally, or ≥38.0°C rectally.
* The primary cause of fever, as determined by the attending physician, is a respiratory tract infection.
* Blood draw is required as part of standard clinical care.
* Ability to comprehend the study's purpose, procedures, and potential risks, and willingness to provide written informed consent.

Exclusion Criteria:

* Inability to provide independent informed consent due to impaired consciousness or other reasons.
* Inability to comply with the study procedures.
* Medical contraindications to blood sampling, such as severe coagulopathy (e.g., INR > 3.0, platelet count < 50 × 10⁹/L).
* Diagnosed with a terminal illness (e.g., advanced malignancy, severe multiple organ failure) and a life expectancy of less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to fever clinics with acute respiratory infections, aged 18 years or older, who provide informed consent. Both sexes are eligible. Participants are observed under standard clinical care without intervention
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Hospitalized for Pneumonia | 30 days
  The percentage of patients who require hospitalization due to radiologically confirmed pneumonia within the 30-day follow-up period.

SECONDARY OUTCOMES:
Rate of Symptom Resolution at 24 Hours | 24 hours
  Proportion of participants achieving complete resolution of patient-reported symptoms (e.g., fever, myalgia) at 24 hours after enrollment.
Rate of Symptom Resolution at 7 Days | 7 days
Time to Sustained Symptom Resolution | 30 days
All-cause Mortality Rate at 30 Days | 30 days
Intensive Care Unit (ICU) Admission Rate at 30 Days | 30 days
Change in White Blood Cell (WBC) Count | Baseline, Day 3
Normalization Rate of C-reactive Protein (CRP) | Baseline, Day 7
Change in Procalcitonin (PCT) Level | Baseline, Day 3
Incidence of Acute Exacerbation of Underlying Chronic Diseases | 30 days
Rate of Unplanned Medical Visits | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
This is an observational real-world cohort study of patients presenting to fever clinics. Individual participant data (IPD) will not be shared because the dataset contains sensitive personal health information, including demographics, clinical findings, and follow-up details. Data privacy and confidentiality will be strictly maintained in accordance with institutional and ethical guidelines.